CLINICAL TRIAL: NCT06099769
Title: A RANDOMIZED, PHASE II STUDY OF ENZALUTAMIDE, ENZALUTAMIDE WITH MIFEPRISTONE, and TREATMENT OF PHYSICIAN'S CHOICE IN PATIENTS WITH AR+ METASTATIC TRIPLE-NEGATIVE OR ER-LOW BREAST CANCER
Brief Title: A Study of Enzalutamide, Enzalutamide in Combination With Mifepristone, or Chemotherapy in People With Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Astellas Pharma US, Inc. (Industry); Breast Cancer Research Foundation (Other); Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 22-334
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer
Keywords: Enzalutamide; Mifepristone; Carboplatin; Paclitaxel; Capecitabine; Eribulin; Triple-negative; Androgen receptor positive; 22-334
MeSH Terms: conditions — Breast Neoplasms | interventions — enzalutamide; Mifepristone

STUDY DESIGN:
Intervention Model Description: This phase II study will randomize.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Enzalutamide (Experimental): Enzalutamide 160 mg/day, continuous daily dosing in a 21-day cycle
  Interventions: Drug: Enzalutamide
- Enzalutamide with Mifepristone (Experimental): Enzalutamide 120mg/day and mifepristone 300mg/day, continuous daily dosing in a 21-day cycle
  Interventions: Drug: Enzalutamide; Drug: Mifepristone
- Chemotherapy:Carboplatin, Paclitaxel, Eribulin or Capecitabine (TPC) (Active Comparator): The treating physician must select from one of the following regimens.
  * Eribulin 1.4 mg/m2 IV Day 1 and Day 8 in a 21-day cycle
  * Capecitabine 1000-1250 mg/m2 twice daily, orally Day 1-14 in a 21-day cycle
  * Paclitaxel 80 mg/m2 IV Day 1, Day 8 in a 21-day cycle
  * Carboplatin AUC 6 IV Day 1 in a 21-day cycle
  * Carboplatin AUC 2 IV Day 1, Day 8 and Day 15 in a 21-day cycle
  Patients randomized to TPC may be offered crossover to enzalutamide plus mifepristone treatment at the time of disease progression if they continue to meet eligibility criteria.
  Interventions: Drug: TPC

INTERVENTIONS:
Drug: Enzalutamide — mouth once daily (160 mg/day)
  Arms: Enzalutamide; Enzalutamide with Mifepristone
Drug: Mifepristone — mouth once daily 300-mg tablet
  Arms: Enzalutamide with Mifepristone
Drug: TPC — The treating physician must select from one of the following regimens:
  * Eribulin 1.4 mg/m2 IV Day 1 and Day 8 in a 21-day cycle
  * Capecitabine 1000-1250 mg/m2 twice daily, orally Day 1-14 in a 21-day cycle
  * Paclitaxel 80 mg/m2 IV Day 1, Day 8 in a 21-day cycle
  * Carboplatin AUC 6 IV Day 1 in a 21-day cycle
  * Carboplatin AUC 2 IV Day 1, Day 8 and Day 15 in a 21-day cycle
  Arms: Chemotherapy:Carboplatin, Paclitaxel, Eribulin or Capecitabine (TPC)

SUMMARY:
The researchers are doing this study to find out if the study drug, enzalutamide, alone or combined with the study drug, mifepristone, is effective in treating advanced or metastatic androgen receptor-positive (AR+) triple negative breast cancer (TNBC) or estrogen receptor-low breast cancer (ER-low BC), and whether these study treatments work as well as standard chemotherapy with carboplatin, paclitaxel, capecitabine, or eribulin.

ELIGIBILITY:
Inclusion Criteria:

Screening Cohort (non-MSK patients only):

* Age ≥18 years at time of consent
* signed the pre-screening informed consent document to allow for AR testing as part of study screening

Treatment Cohort:

* Female or male
* Pathologically confirmed invasive breast cancer that is unresectable, locally advanced, or metastatic
* TNBC (ER/PgR <1%) or ER-low defined as:

  * ER and PgR 1-10%
  * HER2 negative per American Society of Clinical Oncology/College of American Pathologists guidelines
  * Local testing for ER/PgR and HER2 is acceptable for eligibility.
* Tumor must be AR positive. AR is considered positive by IHC if ≥10% of cell nuclei are immunoreactive.

  °AR testing performed locally must use protocol specified methodology to be acceptable for eligibility. Central testing is an option for those unable to perform local testing per this methodology. Please refer to the Section entitled "Treatment Plan" for AR testing methodology or refer to the laboratory manual.
* Evaluable or measurable disease per RECIST version 1.1; subjects with no evaluable AND no measurable disease (e.g., malignant effusions or bone marrow as the only manifestations of disease) are not eligible for enrollment.
* Eligible for one of the chemotherapy options listed as TPC (eribulin, capecitabine, paclitaxel, or carboplatin), as per investigator assessment.
* A representative, formalin-fixed, paraffin-embedded tumor specimen that enables the diagnosis of breast cancer, with adequate viable tumor cells in a tissue block (preferred) or 15 freshly cut unstained slides and 1 H&E slide. Tissue from a metastatic site is preferred.

If not available, tissue from the primary site may be obtained.

* Patients may have received up to 2 prior lines of chemotherapy for metastatic breast cancer.

  * Patients with ER-low breast cancer may receive any number of lines of endocrine therapy +/- targeted therapy (i.e., CDK4/6 inhibitors, PI3K inhibitors).
  * Patients with PD-L1 positive breast cancer (CPS ≥ 10) should have received prior treatment with a checkpoint inhibitor setting unless there is a contraindication to checkpoint inhibitor therapy.
* Patients may receive bisphosphonate or denosumab.
* ECOG performance status 0-2.
* Age ≥18 years.
* Able to understand and the willingness to provide informed consent.
* Patients must not have another active malignancy that requires treatment.
* Women of child-bearing potential and men must agree to use 2 forms of adequate contraception (i.e., barrier contraception, abstinence, intrauterine device, or sterilization method) during study period and for 7 months following treatment end. Women must not breast feed while on study and for at least 3 months after final drug administration.
* Ability to swallow intact enzalutamide and mifepristone.
* Patient must be recovered from any recent major surgery. Radiation must have completed 14 days prior to study start. If treated in the second-line setting, the last chemotherapy or investigational anticancer therapy dose must be at least 14 days prior.
* Adequate organ and marrow function, as defined below:

  * ANC ≥1000, hemoglobin ≥9 g/dL, platelets ≥100,000
  * Total bilirubin ≤1.5x upper limit of normal (ULN), except for patients with known Gilbert syndrome; AST/ALT ≤3x ULN (≤5x ULN if liver metastases); creatinine ≤ 1.5x ULN.
  * Cortisol within normal limits
* Patients must agree to research biopsy at study entry until 40 patients randomized to Arm A and 40 patients randomized to Arm B and 20 patients randomized to Arm C have been biopsied.

  * Biopsy requirement may be waived in consultation with the study PI (Drs. Traina or Nanda) if not medically feasible.

Exclusion Criteria:

* Seizure disorder or any condition that may predispose to seizure (e.g., prior cortical stroke, significant brain trauma) at any time in the past. History of loss of consciousness or transient ischemic attack within 12 months.
* History of brain metastases or leptomeningeal disease.
* Prior antiandrogen therapy (AR antagonist or CYP17 inhibitors).
* Other concurrent investigational anticancer agents.
* Confirmed QT interval with Fridericia correction (QTcF) > 480 msec.
* Any severe concurrent disease, infection, or comorbid condition that renders the patient inappropriate for enrollment in the opinion of the investigator or that interferes with the patient's ability to participate in the study requirements.
* Pregnant patients are not eligible for study.
* Women with a history of unexplained vaginal bleeding or with endometrial hyperplasia with atypia or endometrial carcinoma are excluded from study.
* An active gastrointestinal disorder affecting absorption (e.g., gastrectomy, uncontrolled celiac disease).
* Use of concurrent or chronic daily corticosteroid use. Topical or inhaled corticosteroids are permitted.
* Use of concurrent medications that are strong inducers/inhibitors or substrates of CYP3A4. Patients may be switched to alternative medications for eligibility purposes. A list of CYP3A4 substrates, inducers, and/or inhibitors
* Hypersensitivity reaction to the active pharmaceutical ingredient or any of the tablet components, including Labrasol, butylated hydroxyanisole, and butylated hydroxytoluene.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 2 years
  Response and progression will be evaluated in this study using the international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) Committee (version 1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Traina, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (12):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Francisco (Data collection only), San Francisco, California
  - University of Chicago Medical Center, Chicago, Illinois
  - Dana Farber Cancer Institute (Data Collection Only), Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm